CLINICAL TRIAL: NCT02275546
Title: A Multicenter, Open Label, Randomized, Two-period Crossover Study on the Insertion of MK-8342A (NuvaRing®) Placebo With and Without the Use of NuvaRing Applicator in Healthy Female Subjects
Brief Title: Performance and Safety of Vaginal Ring Applicator in Healthy Females (MK-8342A-063)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 8342A-063
Record Dates: First submitted 2014-10-23; First posted 2014-10-27 (Estimated); Results first posted 2016-04-28 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2022-02

CONDITIONS: Contraception: Optional Applicator for Insertion of Vaginal Ring
MeSH Terms: interventions — NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Applicator→No Applicator (manual) (Experimental): Treatment period 1: Participants will use applicator to insert vaginal ring. Treatment period 2: Participants will manually insert vaginal ring using fingers only.
  Interventions: Drug: Placebo vaginal ring; Device: Single-use, non-sterile applicator
- No applicator (manual)→Applicator (Experimental): Treatment period 1: Participants will manually insert vaginal ring using fingers only. Treatment period 2: Participants will use applicator to insert vaginal ring.
  Interventions: Drug: Placebo vaginal ring; Device: Single-use, non-sterile applicator

INTERVENTIONS:
Drug: Placebo vaginal ring — Drug-free placebo vaginal ring
  Other Names: NuvaRing
Device: Single-use, non-sterile applicator — Single-use, non-sterile, plastic applicator for insertion of vaginal ring.
  Other Names: NuvaRing Applicator

SUMMARY:
The purpose of the study is to assess the performance and safe use of the vaginal ring applicator as an optional aid for insertion of a placebo vaginal ring into the vagina in healthy women

ELIGIBILITY:
Inclusion Criteria:

* healthy, non-pregnant, pre-menopausal female who is not using NuvaRing.
* must meet one of the two following criteria: 1) has not taken a combined hormonal contraceptives for at least 3 months prior to screening and has normal predictable menstrual cycles ranging from 26 to 35 days in length with no history of intermenstrual bleeding in the past 6 months; or 2) has been taking a combined hormonal contraceptive for >3 months and has not experienced unscheduled bleeding for the past 3 months.
* willing to abstain from vaginal penetration, including during sexual intercourse and masturbation, from the time of randomization (Visit 2) to the end of the follow-up period.
* willing to abstain from vaginal penetration with any objects other than the applicator and placebo rings (including but not limited to tampons, douching, use of vaginal applicators for medication, medication, diaphragms, cervical caps, male and female condoms, lubricants, sex toys) from the time of randomization (Visit 2) to the end of the follow-up period.
* good physical and mental health, based upon the medical judgment of the investigator.

Exclusion Criteria:

* current use or has used within past 3 months any of the following: NuvaRing, progestin-only contraceptives (including pills, injection, or implant), oral or transdermal combined hormonal contraceptives with extended or continuous hormonal regimens that prevent monthly withdrawal bleeding by omitting monthly progestin-free intervals. Note: Current use of oral or transdermal combined hormonal contraceptives with 4 to 7 progestin-free days per 28-day cycle for >3 months is permitted.
* has stopped use of any hormonal contraceptive, including NuvaRing, <3 months prior to screening; previous use (≥3 months prior to screening) is permitted.
* history of difficulty retaining NuvaRing in the vagina and therefore could not continue on it as a contraceptive method or difficulty retaining other products (e.g., tampons) in the vagina.
* is pregnant or within 2 months of last pregnancy outcome (delivery, spontaneous or induced abortion, medical or surgical management of ectopic pregnancy).
* is breastfeeding.
* diagnosed or treated for a sexually transmitted disease within the past 6 months.
* current complaints of vaginal or vulvar irritation, discomfort, abnormal bleeding/spotting, or abnormal discharge.
* abnormal cervical Pap smear documented within 12 months of screening.
* genital herpes outbreak in the past 3 years.
* has received any investigational drug or device in the 30 days prior to screening and/or plans to receive any investigational drug or device at any time up to the last protocol-required visit.
* known current gynecological disorder which, in the opinion of the investigator, interferes with the objectives of the study.
* known allergy/sensitivity or contraindication to the investigational product (applicator) or ethylene vinyl acetate.
* current or recent history (within the last six months) of drug or alcohol abuse or dependence.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 164 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2015-04-10 (Actual); Study Completion 2015-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Feldman R, Frenkl TL, Yacik C, Wang Y, Fox MC. Safety and efficacy of the NuvaRing(R) Applicator in healthy females: a multicenter, open-label, randomized, 2-period crossover study. Contraception. 2016 Oct;94(4):362-5. doi: 10.1016/j.contraception.2016.04.017. Epub 2016 May 17. PMID 27207028

RESULTS

PARTICIPANT FLOW:
Groups:
- Applicator→No Applicator (Manual): In Treatment Period 1, participants used the applicator to insert the vaginal ring. In Treatment Period 2 participants manually inserted the vaginal ring using their fingers only.
- No Applicator (Manual)→Applicator: In Treatment Period 1, participants manually inserted the vaginal ring using their fingers only. In Treatment Period 2, participants used the applicator to insert the vaginal ring.
Period: Treatment Period 1
Arm/Group | Applicator→No Applicator (Manual) | No Applicator (Manual)→Applicator
Started | 81 | 83
Completed | 81 | 83
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Applicator→No Applicator (Manual) | No Applicator (Manual)→Applicator
Started | 81 | 83
Completed | 79 | 81
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 164
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.2 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Successful Ring Insertion
Description: Participants completed a Post-Insertion Questionnaire in which they were asked about their experience inserting the vaginal ring. Their answers were recorded and evaluated.
Time Frame: Day 1 (immediately after vaginal ring insertion)
Population: Per Protocol Population, which excluded participants due to important deviations from the protocol that could have substantially affected the results of the efficacy endpoints.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Applicator: Participants used the applicator to insert the vaginal ring.
- No Applicator (Manual): Participants manually inserted the vaginal ring using their fingers only.
Arm/Group | Applicator | No Applicator (Manual)
Number analyzed (Participants) | 102 | 102
Percentage of participants | 100 [96.4 to 100.0] | 100 [96.6 to 100.0]

2. Primary Outcome: Percentage of Participants With Vaginal Ring Expulsion Within 48 Hours of Insertion
Description: Participants completed a Follow-Up Questionnaire in which they asked if they experienced vaginal ring expulsion. Their answers were recorded and evaluated.
Time Frame: Up to 48 hours after vaginal ring insertion
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Applicator | No Applicator (Manual)
Number analyzed (Participants) | 102 | 102
Percentage of participants | 0 [0.0 to 3.6] | 0 [0.0 to 3.6]

ADVERSE EVENTS:
Time Frame: Up to 96 hours after vaginal ring insertion
Description: The safety analysis was based on the All Subjects as Treated (ASaT) Population, which consisted of all randomized participants who attempted to insert a vaginal ring in Treatment Period 1.
Arm/Group | Applicator | No Applicator (Manual)
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/162
Other Adverse Events (participants affected / at risk) | 0/163 | 0/162

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.